CLINICAL TRIAL: NCT03916887
Title: Golf Intervention for Healthy Aging Study
Brief Title: Golf for Healthy Aging
Acronym: GHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Royal & Ancient Group (Unknown)
Responsible Party: Principal Investigator, George Salem, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-17-00004
Record Dates: First submitted 2019-04-04; First posted 2019-04-16 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Exercise Training
Keywords: aging, exercise golf senior intervention

STUDY DESIGN:
Intervention Model Description: Pre-post intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- golf training (Experimental): 10-week golf training program
  Interventions: Behavioral: Golf instruction

INTERVENTIONS:
Behavioral: Golf instruction — Non-golfers instructed to golf over 10 weeks

SUMMARY:
Aging is associated with physiological declines that could impair the ability to perform activities of daily living and thus impair the quality of life of older adults. Golf is an activity that challenges the balance, flexibility, and muscular systems of the golfer and could have important implications in addressing the physiological declines associated with aging. Golf also challenges the cognition of golfer and is typically performed in groups of 2-4 people; therefore, it could also have important implications for the cognitive and social health of older adults. This research will investigate the effects of an introductory, therapeutic golf program on the physiological, cognitive, and social well-being of older adults. 25 older adults (60-80 years) will participate in a 10-week introductory golf program specifically designed with older adults in mind. The intervention will be led by Professional Golf Association (PGA) professionals with experience in teaching older adults to golf. In order to assess the effectiveness of the intervention, the functional, physiological, and cognitive abilities of the participants will be evaluated as well as the overall well-being before and after the completion of the golf program. We will also examine the inflammatory response changes associated with the golf program. These adaptations will be evaluated through the use of biomechanical analysis, standardized older adult functional tests, validated surveys and questionnaires, validated cognitive assessments, and analyses of markers of inflammation.

DETAILED DESCRIPTION:
Implementing a ten-week introductory golf intervention designed for older adults will allow us to evaluate the usefulness of golf as a means to promote physical activity and well-being across the lifespan. Golf, while studied from a performance perspective, has not been studied as an intervention to promote physical activity and health in older adults. This study will contribute to our knowledge about the feasibility and effectiveness of golf as a means to promote wellness across the lifespan.

1.3 HYPOTHESIS

It is hypothesized that, following the intervention, the older adults will demonstrate improved functional, cognitive, and physiological abilities. It is also hypothesized that the participants will demonstrate improvements in golf skill.

2.0 OBJECTIVES AND PURPOSE The purpose of this study is to quantify the changes in functional, cognitive,and physiological abilities following a ten-week introductory golf intervention.

2.1 OBJECTIVE 1: Quantify the changes in the functional, cognitive, and physiological abilities of older adults following a 10-week introductory golf intervention.

Hypothesis: Older adults will demonstrate improved functional, cognitiveand physiological abilities following the intervention.

2.2 OBJECTIVE 2: Quantify golf demands and performance including a biomechanical analysis of golf swings, putting and picking up a ball following a 10-week introductory golf intervention.

Hypothesis: The demands of the golf intervention will be similar to or greater than the demands during commonly utilized older adult balance and strengthening exercises.

2.3 OBJECTIVE 3: Evaluate the safety and feasibility of a 10-week introductory golf intervention.

Hypothesis 3A: Adverse events associated with the intervention will be minor and not more frequent than AE's associated with other activity programs in seniors (e.g. GeroFit).

Hypothesis 3B: Adherence to the program will greater than the adherence associated with other activity-intervention programs in seniors (e.g. GeroFit).

3.0 STUDY DESIGN

We propose a longitudinal study design.

5.0 SELECTION AND WITHDRAWAL OF SUBJECTS

Recruitment: Twenty-five older adults will be recruited to participate in the study.

The potential participants will be recruited by flyers, word of mouth and through the USC Institute of Senior Golf Science webpage. Flyers will be placed at various community centers and senior centers in the cities of South Pasadena, Monterey Park, and the surrounding areas. The flyers will also be placed at both the Arroyo Seco and Monterey Park Golf Courses. The flyer will also be placed on the Institute for Senior Golf Science Facebook Page. Dr. George J. Salem, Kiran Kanwar, Hyun Ji Lee, and Jared Moore will be recruiting potential participants.

A flyer containing general study information will be utilized (see Golf for Healthy Aging Flyer). Included on the flyer is the contact information for the study coordinator, Ms. Kiran Kanwar. Participants will also be recruited through the USC Institute of Senior Golf Science webpage located at http://pt.usc.edu/golfscience. The information included on this webpage is also included (see Golf Healthy Aging Website Recruitment Information). Participants will also be recruited using social media (see Facebook Announcement). Finally, participants will be recruited by word of mouth through a designated personal communication script (see Golf for Healthy Aging Recruitment Script).

During recruitment, potential participants will be informed of the inclusion and exclusion criteria through a two-part screening process.

Phone Screen: Screening (see Golf for Healthy Aging Phone Screen) will consist of a series of questionnaires assessing the potential participant's eligibility for the study. During the initial phone screening, the potential participant will complete the Telephone Memory Impairment Screen validated to assess for dementia and Alzheimer's Disease [21]. The telephone screen will also consist of a series of questions regarding both the inclusion and exclusion criteria described in section 5.1.

Medical Clearance: Following the phone screen, all eligible individuals will be sent a medical clearance form to be taken to their primary care physician. This form will describe the physical requirements of the study so the physician can either approve or deny participation in the study. Included with the form is a description of the study details (see Golf for Healthy Aging Study Information Form), a stamped envelope and one self-addressed envelope to Kiran Kanwar, Golf for Healthy Aging Study Coordinator at the Unversity of Southern California. The participants may either bring in or mail the medical clearance form to their physician and once complete the form will either be mailed or faxed to Kiran Kanwar by the potential participant's primary care physician.

Once the medical clearance form is received, it will be reviewed to confirm whether the participant qualifies. Regardless, the potential participant will be contacted to notify him/her of his/her status in the study. If the participant qualifies, a screening consent enrollment appointment at the University of Southern Calfornia MBRL will be scheduled.

The functional assessments include activities that are regularly conducted throughout the day and have been utilized regularly as part of common clinical practice for assessing functional abilities. In more challenging activities, the participants will be appropriately spotted to ensure safety during the test.

The potential risks are as follows:

Functional Assessment: Fatigue (very minimal risk) - Rest will be provided as needed for the participants.

Muscle soreness (minimal risk) - This is no greater than performing normal activities of daily living.

Joint or muscle injury (minimal risk) - This is no greater than performing normal activities of daily living.

Risk of falling (minimal risk) - On the more challenging tasks, participants will be spotted.

Cognitive Assessment: Questionnaires (minimal risk) - Participants will be given the option to skip or stop answering any questions that make them uncomfortable.

Inflammatory Markers: Infection from blood draws (minimal risk) - A licensed phlebotomist will be making the blood draws.

Golf Intervention: Joint or muscle injury (minimal risk) - The participants will be gradually introduced to the activities associated with the sport of golf. Each golf session will include a sport specific warm-up and exercises that prepare the participants for the daily activities. Additionally, the golfers will be supervised by a PGA Professional who specializes in instructing older adults.

Fatigue (very minimal risk) - Participants will also be allowed rest as needed.

Adverse Events: Any unanticipated problem will be recorded via an incident report (see Golf for Healthy Aging Incident Report). Protocols for the USC MBRL have been developed (see USC Adverse Event Protocol). Any serious adverse event will be reported to the Institutional Review Board at the University of Southern California Health Science Campus using the flow chart below.

Continual Safety Monitoring: Researchers will have weekly meetings with the PGA instructors to keep informed about the intervention and participant safety. Additionally, each week, Kiran Kanwar, Dr. George Salem, Jared Moore, or Hyun Ji Lee, will check in with participants according to the Problem Reports and Tracking Problems Protocol.

9.0 CLINICAL AND LABORATORY EVALUATIONS AND STUDY CALENDAR

Duration and Locations: The study from consent enrollment to final data collection will occur over a 12-week period. The study consists of two to four data collection visits to the Jacquelin Perry Musculoskeletal Biomechanics Research Laboratory (MBRL) in the Division of Biokinesiology and Physical Therapy located on the University of Southern California Health Science Campus. Participants will have the option to complete two of their visits (days 2 and 3) at the golf course in a private room.

University of Southern California MBRL Visits Participants will visit the USC MBRL on four separate occasions. Day 1 will occur following the consent enrollment. Data collection at the MBRL will consist of biomechanical analysis, and functional and physiological testing on two of the days and standardized assessments and questionnaires of cognition and self-efficacy, and a blood draw on the other two days.

Biomechanical Analysis (minimal risk): Laboratory kinematics and kinetics will be collecting using an 11-camera digital motion capture system (Qualysis, AB, Gothenberg, Sweden). 14 mm reflective markers will be used to define body segments and track motion during the trials. The trunk will be modeled as 4 rigid segments: pelvic, lumbar, thoracic and head segments. The lower extremity will be modeled as 3 rigid segments: thigh, shank and foot. The upper extremity will be modeled as 3 rigid segments: upper arm, forearm and hand. The trunk will be modeled as 2 rigid segments: upper and lower trunk.

Assessment of Inflammation Markers (blood draw minimal risk):

We will assess the chronic immune response to the golf-training program by examining the inflammation markers C-reactive protein (CRP), interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-a). Older adults show signs of increased low-grade, chronic inflammation by exhibiting higher blood plasma levels of these cytokines (Franceschi & Campisi, 2014). These elevated, sub-clinical levels could cause detriments to physical functionality (such as grip strength), which we will be testing further in our study (Brinkley et al., 2009). Previous reports show that aerobic exercise can help to attenuate these elevated levels in older adults (Colbert et al., 2004; Kohut et al., 2006). We will be examining the effect of a golf-program intervention study on the chronic levels of these cytokines to promote golf as a unique intervention for the maintenance of plasma cytokines and functional ability in older adults.

Fasting (12h) blood will be drawn from the antecubital vein (~20cc) by a licensed phlebotomist at the second baseline and 10-week follow-up visits. Participants will receive refreshment after blood draw and prior to further testing. Plasma will be harvested into 500ul cryovials and stored in -80oC at the Harlyne J. Norris Research Tower (HNRT) on the USC Health Sciences Campus.

Day 1 Tasks (minimal risk): Data collection will last approximately 2 hours and will include previously validated functional assessments.

* Height, mass, resting heart rate, resting blood pressure and body fat percentage via Bioelectrical Impendence Analysis
* Senior Fitness Test: 30 second chair stand, , 6 minute walk test, , heel-rise test, 8 foot-up-and-go test [23].
* Functional Reach Test
* Hip and knee muscle performance testing [24]
* Gait analysis
* Quiet standing (Eyes Open, Eyes Closed, Tandem Standing)
* Balance confidence as assessed by the Activities Specific Balance Confidence (ABC) Scale [26].
* Participants will be given a Golf History Form to complete at home and return on Day 2 of testing at USC.

Day 2 Tasks (minimal risk): Data collection will last approximately 1.5 hours and will include previously validated cognitive and self-efficacy assessments. Participants will have the option to complete this testing day at the golf course in a private room to reduce travel for testing.

* Participants will turn in their Golf History Form
* Self-reported health-related quality of life as assessed by the RAND 12-item Health Survey[27-29]
* Surveys from the Midlife in the United States Survey (MIDUS) study assessing Positive and Negative affect [30], Social Well-Being [31] and Sense of Control [32].
* Cognition as assessed by the NIH Toolbox for cognition [33] using the following scales:

  * Dimensional Change Card Sort Test - Executive function, set-switching
  * Flanker Inhibitory Control and Attention Test - Exexcutive function, visuospatial inhibitory attention
  * List Sorting Working Memory Test - Executive function, working memory
  * Picture Sequence Memory Test - Episodic memory
  * Pattern Comparison Processing Speed Test - Processing speed
* Physical activity habits will be assessed via a questionnaire developed by the Postmenopausal Estrogen/Progestins Intervention (PEPI) Study [34, 35] and a physical activity free recall.
* Episodic verbal learning and memory as assessed by the California Verbal Learning Test.
* Blood draw for assessment of inflammation markers

Day 3 Tasks (minimal risk): This data collection will occur following the 10-week training intervention. Data collection will last approximately 1.5 hours and will include previously validated cognitive and self-efficacy assessments. Participants will have the option to complete this testing day at the golf course in a private room to reduce travel for testing.

* Self-reported health-related quality of life as assessed by the RAND 12-item Health Survey[27-29]
* Surveys from the Midliefe in the United States Survey (MIDUS) study assessing Positive and Negative affect [30], Social Well-Being [31] and Sense of Control [32].
* Cognition as assessed by the NIH Toolbox for cognition [33] using the following scales:

  * Dimensional Change Card Sort Test - Executive function, set-switching
  * Flanker Inhibitory Control and Attention Test - Exexcutive function, visuospatial inhibitory attention
  * List Sorting Working Memory Test - Executive function, working memory
  * Picture Sequence Memory Test - Episodic memory
  * Pattern Comparison Processing Speed Test - Processing speed
* Physical activity habits will be assessed via a questionnaire developed by the Postmenopausal Estrogen/Progestins Intervention (PEPI) Study [34, 35] and a physical activity free recall.
* Episodic verbal learning and memory as assessed by the California Verbal Learning Test.
* Blood draw for assessment of inflammation markers

Day 4 Tasks (minimal risk): This data collection will occur following the 10-week training intervention. Data collection will last approximately 3 hours and will include previously validated functional assessmentsand a series of golf related movements.

* Height, mass, resting heart rate, resting blood pressure and body fat percentage via Bioelectrical Impendence Analysis
* Senior Fitness Test: 30 second chair stand, , 6 minute walk test, , heel-rise test, 8 foot-up-and-go test [23].
* Hip and knee muscle performance testing [24]
* Gait analysis
* Quiet Standing (Eyes Open, Eyes Closed, Tandem standing)
* Balance confidence as assessed by the Activities Specific Balance Confidence (ABC) Scale [26].
* Golf swings, chips and putts that are common to recreational golf players. Participants will perform up to 5-10 trials of each swing type.
* Picking up and setting down a golf ball. Subjects will perform up to 5-10 trials of each strategy.
* Exit questionnaire about golf training program

At 6-months post training, participants will be mailed and asked to complete surveys from the Midlife in the United States Survey (MIDUS) study assessing Positive and Negative affect [30], Social Well-Being [31] and Sense of Control [32]. They will also be mailed the physical activity free recall. These can be mailed to study coordinator, Kiran Kanwar in the included self-addressed and stamped envelopes.

Six months after the completion of the study, participants will receive a telephone call to follow-up on their current golf playing habits following the 10-week program. The telephone survey questions can be found in the Golf Play Telephone Survey.

Analysis: Laboratory-based kinematics, and kinetics will be managed by MATLAB with a custom written code for data processing. The functional assessments and self-reported quality of life will be scored according to standard clinical practice.

Golf Training Visits Participants will participate in golf training programs at the Arroyo Seco Golf Course in South Pasadena or the Monterey Park Golf Club in Monterey Park.

The Arroyo Seco Golf Course is an 18-hole, community golf course located in South Pasadena, CA. During the intervention, golfers will be allowed to play as many or as few holes as desired. The Arroyo Seco Golf Course also has a driving range where participants will be able to practice their swings before progressing to golf play.

The Monterey Park Golf Club is a 9-hole, 3-park golf course (beginner course) located in Monterey Park, CA. During the intervention, golfers will be allowed to play as many or as few holes as desired. The Monterey Park Golf Clib also has a driving range where participants will be able to practice their swings before progressing to golf play.

Participants will be divided into groups of 2-4 golfers and will meet with a PGA Professional two times per week for ten weeks. Training sessions will last 1-2 hours. The program is specifically designed for older adults not currently playing golf. Training will include a warm-up that prepares the participants for the activities to be practiced, flexibility and strengthening exercises to prepare the participants for the golf activities, and a gradual introduction to golf play. The first set of sessions will include introduction to the different forms of the golf swing beginning with partial swings and then gradually progressing to a full swing. Swing modifications will be provided on an individual basis to address needs of the participant. Golf play will begin on holes that are flatter and close to the clubhouse and will begin by only playing 1-2 holes. The golfers will then be appropriately progressed to longer golf play as the PGA Professional feels it is appropriate. All equipment and fees will be included and there will be no cost to the participants.

Tasks (minimal risk):

* Warm-up: Each training session will begin with a sport specific warm-up that prepares the participants for the activities of the day.
* Supplementary Exercises: Additional strengthening and flexibility exercises will be included in training sessions to prepare the participants for golf-related activities.
* Golf swings and putting: These movements will be introduced in a progressive nature beginning with partial swings of the least forceful swing type and eventually progressing to the more forceful swings (drives). Swings with the following equipment will be included: putters, pitching or sand wedges, irons, and woods.
* Picking up a ball: The participants will be introduced to techniques to picking up a golf ball which will be individualized to the needs of the participants based off current research in the MBRL (HS-15-00038).
* Walking: Participants will gradually increase walking distance. Practice will begin on flat holes and will progress to holes with more challenging terrain.
* Golf play: Participants will be gradually introduced to regular golf play beginning with play on a single, low difficulty hole and progressing to multiple holes. Skill difficulty will also be gradually increased.
* During the intervention, walking distance will be tracked via fitness trackers. Golf performance will be tracked as well.

10.0 CRITERIA FOR EVALUATION AND ENDPOINT DEFINITIONS

All subjects will be evaluated on the dependent variables listed in section 13.0.

Endpoint Definitions - not applicable.

11.0 SPECIAL INSTRUCTIONS:

Not applicable

12.0 DATA COLLECTION AND MONITORING

* Motion capture kinetics and kinematics
* Inflammation markers C-reactive protein (CRP), interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-a)
* Functional assessment scores (Tests listed in 9.0)
* Self-reported quality of life (Tests listed in 9.0)
* Sense of control, positive and negative affect, social well-being
* Physical activity recall

Data will be stored securely in the MBRL, CHP, room G9. Electronic data will be stored on a password protected computer. Hard copies of data will be stored in a locking file cabinet. No subject identifiers will be collected.

13.0 STATISTICAL CONSIDERATIONS

13.1 PRIMARY DEPENDENT VARIABLES

13.1.1 Segment and joint angular positions, velocities and accelerations 13.1.2 Joint torques 13.1.3 COP excursion, sway amplitude and velocity 13.1.4 COM excursion 13.1.5 Static and dynamic balance 13.1.6 Hip and Knee Muscle Performance 13.1.7 Gait speed 13.1.8 Gait spatiotemporal characteristics 13.1.9 Cognitive-Motor Dual Task Performance 13.1.10 Activities Specific Balance Confidence 13.1.11 Senior Fitness Test 13.1.12 Self-Rated Health 13.1.13 Verbal memory recall 13.1.14 Positive Affect 13.1.15 Negative Affect 13.1.16 Personal Mastery 13.1.17 Perceived Constraints 13.1.18 Social Contribution 13.1.19 Cognition Fluid Composition Score

13.2 POWER ANALYSIS

To date, this study has not been conducted and thus no preliminary data was available for a power analysis. 25 subjects are requested to ensure for adequate sample size and account for study attrition, based on other exercise intervention studies in older adults [36, 37].

13.3 STATISTICAL ANALYSIS Within subject, pre-intervention and post-intervention comparisons will be made for variables.

14.0 REGISTRATION GUIDELINE

Following confirmation of the inclusion and exclusion criteria, all potential participants will be consented before enrollment in the study. Dr. George J. Salem, Kiran Kanwar, Hyun Ji Lee, and Jared Moorewill be obtaining consent. George J. Salem, Kiran Kanwar, Hyun Ji Lee, and Jared Moore have undergone CITI Training for human subjects' research. In order to participate in the study, participants must be English speaking and have the ability to follow instructions (as assessed by the Telephone Memory Impairment Screen); therefore, there is no need of a legally authorized representative during the consent process. Participants will be consented using a USC Informed Consent form after being explained the details of the study and allowing for adequate time to ask questions and make a decision.

ELIGIBILITY:
Inclusion Criteria:

* • Older adult: 60-80 years old

  * The ability to stand independently without external support
  * No or minimal previous golf experience
  * Played <1 time in the past 6 months
  * Played ≤3 times in the past 2 years
  * English Speaking

Exclusion Criteria:

* • Dementia and Alzheimers Disease assessed via the Telephone Memory Impairment Screen [21]

  * Symptomatic cardiovascular disease, active angina, uncontrolled hypertension (SBP>160 or DBP>90, high resting pulse HR>90), symptomatic orthostatic hypotension
  * Unstable asthma, exacerbated COPD
  * Rheumatoid arthritis, unstable ankle, knee, hip, shoulder or wrist joints
  * History of injury or orthopedic operation within the last 6 months
  * Movement disorders (Parkinson's disease or other neurological disorders), stroke, hemiparesis or paraparesis
  * Peripheral neuropathies, severe vision or hearing problems, or metastatic cancer
  * Individuals with vestibular, visual, musculosketelal, orthopedic and/or neurological disorders known to impair balance

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Change in Gait speed | baseline and after 10 weeks
  change in walking speed

SECONDARY OUTCOMES:
Change in Strength | baseline and after 10 weeks
  change in dynamic and static strength

OTHER OUTCOMES:
Change in Cognition | baseline and after 10 weeks
  change in NIH Cognitive Toolbox scores
Change in Balance | baseline and after 10 weeks
  change in dynamic and static balance

CONTACTS AND LOCATIONS:
Locations (1):
- University Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No